CLINICAL TRIAL: NCT01877135
Title: Malignant Progression of Anal Intra-epithelial Neoplasia in a Cohort of Patients
Acronym: AIN3
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: French Society of Coloproctology (Other)
Collaborators: Société Nationale Française de Gastroentérologie (Other)
Responsible Party: Sponsor
Other Study IDs: 11-LAZ-001
Record Dates: First submitted 2013-06-11; First posted 2013-06-13 (Estimated); Last update posted 2015-03-05 (Estimated); Status verified 2013-09

CONDITIONS: Anal AIN3; Anal Carcinoma
Keywords: anal carcinoma; AIN3; cohort study
MeSH Terms: conditions — Anus Neoplasms

STUDY DESIGN:
Observational Model: Cohort
Biospecimen Retention: Samples Without DNA — A liquid phase anal smear
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Anal AIN3: patients > 18 years, with anal AIN3, without history of anal carcinoma

SUMMARY:
Evaluation of the 3-years anal carcinoma (AC) incidence in patient with anal AIN3 lesions, and factors associated with this AC. A retrospective cohort study will be conducted (2000-2013) followed by a prospective cohort study (starting in 2013) with new diagnoses of anal AIN3 lesion. The main outcome is histology proven AC. The 3-years incidence rate of AC will be calculated. Factors associated with AC will be estimated using a multivariate Cox regression model.

DETAILED DESCRIPTION:
"Background : Incidence of anal carcinoma (AC) is considerably increasing, but no data on risk of AC in patient with anal AIN3 lesions are available, nor french recommendations about screening and treatment of anal AIN3 lesions.

Objective : Evaluation of the AC incidence in patient with anal AIN3 lesions, and factors associated with this AC.

Population : Patients with a diagnosis of anal AIN3 lesion will be included and followed for 3 years. Patients with past history of AC won't be included.

Study design : Retrospective cohort study will be conducted from 2000 using diagnostic codes of anal AIN3 lesion in histo-pathology departments. Then a prospective cohort study will be conducted with new diagnoses of anal AIN3 lesion.

Outcome : The main outcome is histology proven AC. AC identification can be done either by using diagnostic codes of AC in histo-pathology departments (for retrospective cases), or prospectively.

Statistics : The incidence rate of AC will be calculated. Factors associated with AC will be estimated using a multivariate Cox regression model.

Number of patients : 1000 Number of centers : 35 Length of follow-up: 3 years at least Length of study : 3 years of inclusion and 3 years of follow-up at least"

ELIGIBILITY:
Inclusion Criteria:

To be included in the cohort, patients have to:

- have an anal AIN3 (including Bowen's disease) diagnosed by histology (screening population, post-operative discovery…)

* Aposteriori for patients with a history of anal AIN3 complicated or not by an anal cancer. These cases will be identified from data bases of anatomopathology laboratories in hospitals since January 1st 2000.
* At the diagnostic for the new anal AIN3 Units care involved in the study are those involved in the follow-up of patients with anal pathologies en France, especially anal cancer. Samples are analyzed by the laboratories of anatomopathology of the hospitals where the patients are diagnosed. These points make the histological data bases reliable and allow clearly identifying cases of anal ain3 retrospectively since 2000.

Taking in account the number and quality of the units care involved in the study and the way cases are identified, we think our recruitment will be exhaustive in France, to limit selection bias.

- Patient's non opposition to study

Exclusion Criteria:

* history of anal carcinoma without any history of anal AIN3 lesion
* impossible follow-up for the duration of the study (3 years or more)
* patient aged under 18

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients consulting a proctologist in primary care or in hospital
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2013-08; Primary Completion 2016-06 (Estimated); Study Completion 2019-06 (Estimated)

PRIMARY OUTCOMES:
at least one anal cancer | 3-year incidence of anal carcinoma
  the first diagnosis of anal carcinoma

SECONDARY OUTCOMES:
Observance | 3 years
  Observance defined by at least one consult a year, in case of history anal dysplasia, or 2 consults a year, in case of persistence of anal dysplasia
patient's feelings about his therapeutic care and impact on his emotional life | 3 years
  Patient's feelings about his therapeutic care and impact on his emotional life will be evaluated with a single question with an analogical visual scale from 0 (I'm feeling very bad) to 10 (I'm feeling very good)

CONTACTS AND LOCATIONS:
Overall Officials: Laurent Abramowitz, MD, Principal Investigator — Assistance Publique Hopitaux de Paris
Locations (1):
- Service d'Hépato-gastro-entérologie, Hôpital Bichat, 46 rue Henri Huchard, Paris, Paris, France